CLINICAL TRIAL: NCT04428177
Title: Intravascular Lithotripsy in the Treatment of Calcified Coronary Lesions - Coronary Calcification Study
Brief Title: Coronary Calcification Study - Intravascular Lithotripsy for Calcified Lesions
Acronym: CCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/RVO-FNOs/2020
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Calcification
Keywords: Coronary Artery Calcification; Intravascular Lithotripsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrvascular Lithotripsy (Experimental): Calcified coronary lesions will be treated with intrvascular lithotripsy
  Interventions: Device: Intravascular lithotripsy
- Standard therapy (Active Comparator): Standard treatment of calcified coronary lesions: cutting, scoring or non-compliant balloon predilatation or rotational atherectomy
  Interventions: Device: Standart therapy

INTERVENTIONS:
Device: Intravascular lithotripsy — Intravascular lithotripsy uses sonic pressure waves to disrupt calcium with minimal impact to soft tissue of coronary vessel
  Arms: Intrvascular Lithotripsy
Device: Standart therapy — conventional preparation of calcified lesion: non-compliant, cutting or scoring ballons predilatation or rotational atherectomy
  Arms: Standard therapy

SUMMARY:
The aim of this prospective randomised study is to compare the safety and efficacy of novel intravascular lithotripsy (IVL) to the standard therapy of calcified coronary lesions.

DETAILED DESCRIPTION:
The study will include a total of 40 patients with calcified coronary lesions who will be randomised 1:1 to the treatment with IVL (Shockwave; Shockwave Medical, Inc, Santa Clara, USA) or the standard therapy (non-compliat high-pressure or Scoreflex predilatation, rotational atherectomy, etc). Appropriate preparation of the lesions will be followed by DES implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed, written consent by the patient
* Ability to comply fully with the study protocol
* Negative pregnancy test (and effective contraception) in women with childbearing potential

Angiographic inclusion criteria:

* Native coronary artery lesion with diameter stenosis ≥50% suitable for PCI
* Heavy calcification, defined as calcification within the lesion on both sides of the vessel assessed during angiography
* Reference vessel diameter (RVD) ≥2.5 mm with lesion length <32 mm
* TIMI flow 3 of the target vessel at baseline
* No visible thrombus at target lesion site

Exclusion Criteria:

* Cardiogenic shock or haemodynamic instability requiring mechanical circulatory support
* Active malignancy or other comorbidities with a life expectancy of 12 months
* Limited the possibility of control coronaro angiography (e.g., advanced renal failure)
* Known allergy to contrast agents (that cannot be adequately premedicated) or required concomitant dual antiplatelet therapy
* Current problems with substance abuse (e.g., alcohol or drugs)
* Subject is participating in another investigational drug or device clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal lumen diamether (MLD) | 1 year
  minimal diamether of treated lesion measured by quantitative coronary angiography
Late luemn loss (LLL) | 1 year
  difference between post-procedure MLD and 12-month MLD

SECONDARY OUTCOMES:
Binary in-stent restenosis | 1 year
  diamether stenosis ≥ 50% of reference vessel
Major adverse cardiac events (MACE) | 1 year
  Cardiac death, myocardial infarction or tagret lesion revascularisation (TVR)

OTHER OUTCOMES:
Angiographic success | up to end of the procedure, an average of 2 hours
  success in facilitating stent delivery with <50% residual stenosis and without serious angiographic complications
Clinical success | up to discharge, an average of 3 days
  angiographic success with no evidence of in-hospital MACE

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Diseases, University Hospital, Ostrava, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pleva L, Kukla P, Konde A. Comparison of the efficacy of intravascular lithotripsy and rotational atherectomy as adjunctive therapy before drug-eluting stent implantation in calcified coronary lesions (CCS- Coronary Calcification Study). BMC Cardiovasc Disord. 2025 Sep 2;25(1):648. doi: 10.1186/s12872-025-05082-z. PMID 40898049